CLINICAL TRIAL: NCT05528289
Title: Effects on PaCO2 Levels of Two Different Nasal Cannula in COPD Patients With Persistent Hypercapnia Following an Acute Severe Exacerbation
Brief Title: Effects on PaCO2 Levels of Two Different Nasal Cannula in COPD Patients
Acronym: CODUET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: n° 174/2022/Disp/AOUBo
Record Dates: First submitted 2022-08-09; First posted 2022-09-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: HFNC; Hypercapnia; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC 40 L/min with conventional symmetric nasal cannula (Active Comparator): The patients will be asked to breathe with HFNC at flow of 40 L/min with standard interface
  Interventions: Device: AIRVO 2, the new asymmetric nasal cannula
- HFNC 40 L/min with new asymmetric nasal cannula (Active Comparator): The patients will be asked to breathe with HFNC at flow of 40 L/min with the new asymmetric nasal cannula
  Interventions: Device: AIRVO 2, with conventional symmetric nasal cannula

INTERVENTIONS:
Device: AIRVO 2, with conventional symmetric nasal cannula — The patients will be asked to breathe with HFNC at flow of 40 L/min with the standard cannula
  The size of nasal cannula will be selected to occlude patient's nostril of about 2/3.
  Temperature will be set according to the patient's tolerance starting from 31°C, up to 37°C, while FiO2 is adjusted to maintain SpO2 between 88 and 92%.
  Other Names: standard cannula
  Arms: HFNC 40 L/min with new asymmetric nasal cannula
Device: AIRVO 2, the new asymmetric nasal cannula — The patients will be asked to breathe with HFNC at flow of 40 L/min with the new asymmetric nasal cannula
  The size of nasal cannula will be selected to occlude patient's nostril of about 2/3.
  Temperature will be set according to the patient's tolerance starting from 31°C, up to 37°C, while FiO2 is adjusted to maintain SpO2 between 88 and 92%.
  Other Names: "Optiflow+ Duet"
  Arms: HFNC 40 L/min with conventional symmetric nasal cannula

SUMMARY:
High-flow nasal cannula (HFNC) therapy is increasingly used in the management of acute respiratory failure. Its clinical application has been expanded also in other specific settings In stable COPD patients and in those recovering from acute exacerbation, HFNC can reduce PaCO2, respiratory rate, minute ventilation and respiratory effort.

The aim of this randomized crossover physiological study is to investigate the effects on PaCO2 levels of two different nasal cannula ('Optiflow + Duet' interface vs "standard" nasal interface) in COPD patients with persistent hypercapnia following an acute severe exacerbation

ELIGIBILITY:
Inclusion Criteria:

* Inpatients recovering from an acute exacerbation of their disease
* Persisting hypercapnia, despite having reached a stabilization in pH (i.e. pH>7,35 and
* PaCO2>50 mmHg on 3 consecutive measurements)
* Informed consent

Exclusion Criteria:

* Body Mass Index (BMI) > 30 kg/m2;
* Previous diagnosis of Obstructive sleep apnea syndrome (OSAS)
* Chest wall disease
* Heart failure
* Severe hemodynamic instability ( need for amine support)
* Acute coronary syndrome (ACS)
* Severe arrhythmia
* Renal insufficiency
* Patients unable to protect respiratory airways
* Respiratory arrest and need for endotracheal intubation
* Pregnancy
* Need for sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changes of the partial pressure of carbon dioxide (PaCO2) levels | immediately after intervention
  Arterial Blood Gases will be analyzed from a sample taken from the arterial artery

SECONDARY OUTCOMES:
Respiratory Rate ( RR), (b/min) | 90 minutes
  This parameter will be measured by a bioelectrical impedance monitor and a single-use Pad Set sensor that will be placed on the surface of the chest wall (ExSpiron, Respiratory Motion) Inc. USA)
Tidal Volume ( TV), (mL) | 90 minutes
  This parameter will be measured by a bioelectrical impedance monitor and a single-use Pad Set sensor that will be placed on the surface of the chest wall (ExSpiron, Respiratory Motion) Inc. USA)
Minute Ventilation (VE), (L/min) | 90 minutes
  This parameter will be measured by a bioelectrical impedance monitor and a single-use Pad Set sensor that will be placed on the surface of the chest wall (ExSpiron, Respiratory Motion) Inc. USA)
Inspiratory effort quantification | 90 minutes
  Esophageal pressure assessment through dedicated esophageal pressure transducer ( (Marquat Genie Biomedical,France)
Transcutaneous carbon dioxide (TcPCO2) and oxygen saturation (SpO2) | 90 minutes
  TcPCO2 and SpO2 will be recorded by using a dedicated device (SenTec AG, Therwil, Switzerland)
Dyspnea score | immediately after intervention
  Dyspnea will be recorded using the Borg scale that is a numeric scale where 0 is no dyspnea and 10 the maximal dyspnea that a patient can imagine
Comfort | immediately after intervention
  this will be assessed by using the Visual Numerical Scale ranging between 1 (extreme discomfort) and 5 (very comfortable),

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico di Sant'Orsola, Bologna, Italy